CLINICAL TRIAL: NCT06109571
Title: Clinic-level Implementation of mHealth to Improve HIV Viral Suppression for Patients With Substance Use Disorders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-0938; 1R01DA055527-01A1 (NIH); Protocol Version 11/14/2024 (Other: UW Madison); A534265 (Other: UW Madison); SMPH/MEDICINE/INFECT DIS (Other: UW Madison)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Substance Use Disorders
Keywords: Viral Suppression; mHealth
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Stepped-wedge, one-way crossover, cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Group 1: mHealth Implementation (Experimental): First 2 sites begin enrollment. Research participants will be asked to complete weekly-check-in, 4 research surveys and engage in content available in the Connections app and with peer mentors over the course of a year.
  Interventions: Device: Connections App
- Group 2: mHealth Implementation (Experimental): Next 2 sites begin enrollment 6 months after Group 1. Research participants will be asked to complete weekly-check-in, 4 research surveys and engage in content available in the Connections app and with peer mentors over the course of a year.
  Interventions: Device: Connections App
- Group 3: mHealth Implementation (Experimental): Next 2 sites begin enrollment 6 months after Group 2. Research participants will be asked to complete weekly-check-in, 4 research surveys and engage in content available in the Connections app and with peer mentors over the course of a year.
  Interventions: Device: Connections App
- Group 4: mHealth Implementation (Experimental): Next 2 sites begin enrollment 6 months after Group 3. Research participants will be asked to complete weekly-check-in, 4 research surveys and engage in content available in the Connections app and with peer mentors over the course of a year.
  Interventions: Device: Connections App

INTERVENTIONS:
Device: Connections App — The Connections app was developed for patients with substance use disorders or unhealthy substance use and adapted to include HIV support. For this study, it has been modified to provide additional resources to support patients engaged in HIV care. Connections' core features include agency-specific informational resources compiled in a resource center, patient self-monitoring through weekly check-in surveys, discussion rooms, and private messaging.

SUMMARY:
The current protocol aims to enroll up to 806 participants from 8 study sites in a clinic-supported intervention which will connect them to Vivent Health care team and a cohort of peer mentors for a year-long intervention period to support patient HIV care to maintain viral suppression and clinic appointments.

DETAILED DESCRIPTION:
This protocol describes the implementation phase of a 5-year NIH-funded research project designed to evaluate the effectiveness of an innovative clinic-level intervention featuring an evidence-based, HIPAA-compliant mobile health (mHealth) application ("Connections," a smartphone app operated by the company CHESS Health) and peer-driven social support.

The goal of this project is to implement and evaluate an evidence-based mHealth system to improve HIV viral suppression and reduce missed clinic visits within a multi-site, comprehensive HIV care program. Connections is a mobile health app developed by CHESS Health to support patients with substance use disorders.

The investigators hypothesize that implementation of an adapted version of Connections within an established network of HIV clinical practices will reduce the occurrence of the primary outcome of virologic failure and the secondary outcome of missed clinic appointments.

The specific aims are:

1. To test the effectiveness of Connections using a stepped-wedge randomized trial.
2. To evaluate the implementation of Connections within the HIV Medical Home Model. Using the RE-AIM framework, we will analyze patient-level, provider-level, and clinic-level factors that influence the reach, implementation, adoption, and maintenance of Connections in HIV practices.
3. To systematically measure costs of implementation of Connections in relationship to its benefits related to preventing virologic failure and missed clinic appointments.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write and speak English
* Receives HIV Disease Care at Vivent Health
* At risk for poor engagement in HIV care, as evidenced by any one of the following:

  * Prior missed clinic visits
  * Poor adherence to medical treatment defined as 2 or more missed doses of medication in a month
  * Unhealthy alcohol or other substance use, as evidenced by a diagnosis of substance use disorder on the patient's problem list, a prior referral to alcohol or substance abuse services, or answering "yes" to one or both of the following screening questions:

    * Has drinking alcohol or using drugs (including marijuana) ever caused problems in your life, such as damaging relationships, causing you to not meet obligations at work, or getting in trouble with the law?
    * Are you currently participating in any treatment or counseling because of problems caused by drug use? This can include groups like N. A., or one-on-one interaction with a doctor or therapist.

Exclusion Criteria:

* Individuals who do not currently have a smartphone or are unwilling to obtain a smartphone will not be able to participate in this study.
* People who are unwilling to download and activate the Connections app.
* People with cognitive or other impairment that precludes the capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Virologic Failure | baseline and 12 months for each clinic
  Using the stepped-wedge design to assess Effectiveness, each site will function as its own control or "usual care" group prior to implementation of Connections. (Aim 1)
Percentage of Vivent Health HIV patients who have downloaded and used Connections | up to 4 years
  The primary Reach measure will be the percentage of Vivent Health HIV patients who have downloaded and used Connections, including sex, racial, and ethnic characteristics. (Aim 2)
Incremental Cost per Quality-Adjusted Life-Year Gained through Increased Antiretroviral Adherence | up to 12 months
  Setup, operating, and healthcare costs of implementation in relationship to its effectiveness in preventing virologic failure and missed clinic appointments. The primary incremental cost-effectiveness ratio (ICER) will be the incremental cost per quality-adjusted life-year gained through increased antiretroviral adherence (Aim 3)

SECONDARY OUTCOMES:
Number of Missed Clinic Appointments | baseline and 12 months for each clinic
  Using the stepped-wedge design to assess Effectiveness, each site will function as its own control or "usual care" group prior to implementation of Connections. (Aim 1)
Number of "meaningful use" weeks | up to 12 months
  Adoption at the patient level is based on research-driven metrics of "meaningful use" for mHealth, defined as a patient accessing any part of Connections beyond the home page during a given week in the 12-month period after downloading the app. (Aim 2)
Days of "meaningful use" per week | up to 12 months
  Adoption at the patient level is based on research-driven metrics of "meaningful use" for mHealth, defined as a patient accessing any part of Connections beyond the home page during a given week in the 12-month period after downloading the app. (Aim 2)
Change in "meaningful use" after a private message | before and after messaging (any time up to 12 months)
  The investigators will assess whether receiving a message through Connections (for example, a private message from a case manager after a missed appointment) is associated with subsequent patient use of Connections. (Aim 2)
Percent Participant Follow up in the 6-month post-intervention period | clinic follow up in the 6-month post-intervention period (up to 18 months for participant)
  Maintenance is defined as follow up on the effectiveness measures (viral load and missing-visit rates) in the 6-month post-intervention period. (Aim 2)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Westergaard, Principal Investigator — UW School of Medicine and Public Health; Andrew Quanbeck, Principal Investigator — UW School of Medicine and Public Health
Locations (8):
- United States (8):
  - Vivent Health Clinic, Denver, Colorado
  - Vivent Health Clinic, Kansas City, Missouri
  - Vivent Health Clinic, St Louis, Missouri
  - Vivent Health Clinic, Austin, Texas
  - Vivent Health Clinic, Green Bay, Wisconsin
  - Vivent Health Clinic, Kenosha, Wisconsin
  - Vivent Health Clinic, Madison, Wisconsin
  - Vivent Health Clinic, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF